CLINICAL TRIAL: NCT04124484
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of DBPR108 Tablets for Type 2 Diabetes Mellitus
Brief Title: DBPR108 Tablets in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPC/HA1117/PRO-II
Record Dates: First submitted 2019-07-08; First posted 2019-10-11 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DBPR108; type 2 diabetes mellitus; DPP4 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — DBPR108

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 50mg group (Experimental): Participants received one 50mg of DBPR108 tablet and two placebos matching DBPR108 100mg under fasted conditions for one day.
  Interventions: Drug: DBPR108 tablet(50mg), Placebo matching DBPR108 tablet(100mg)
- 100mg group (Experimental): Participants received one 100mg of DBPR108 tablet and two placebos matching DBPR108 50mg and 100mg under fasted conditions for one day.
  Interventions: Drug: DBPR108 tablet(100mg), Placebo matching DBPR108 tablet(50mg), Placebo matching DBPR108 tablet(100mg)
- 200mg group (Experimental): Participants received two 100mg of DBPR108 tablets and one placebo matching DBPR108 50mg under fasted conditions for one day.
  Interventions: Drug: DBPR108 tablet(100mg), Placebo matching DBPR108 tablet(50mg)
- placebo group (Placebo Comparator): Participants received two placebo matching DBPR108 100mg and one placebo matching DBPR108 50mg
  Interventions: Drug: Placebo matching DBPR108 tablet(100mg), Placebo matching DBPR108 tablet(50mg)

INTERVENTIONS:
Drug: DBPR108 tablet(50mg), Placebo matching DBPR108 tablet(100mg) — One DBPR108 tablet(50mg) administered orally once a day + Two Placebos matching DBPR108 tablet(100mg) administered orally once a day for 12 weeks
  Arms: 50mg group
Drug: DBPR108 tablet(100mg), Placebo matching DBPR108 tablet(50mg), Placebo matching DBPR108 tablet(100mg) — One DBPR108 tablet(100mg) administered orally once a day + One Placebo matching DBPR108 tablet(100mg) administered orally once a day + One Placebo matching DBPR108 tablet(50mg) administered orally once a day for 12 weeks
  Arms: 100mg group
Drug: DBPR108 tablet(100mg), Placebo matching DBPR108 tablet(50mg) — Two DBPR108 tablets(100mg) administered orally once a day + One Placebo matching DBPR108 tablet(50mg) administered orally once a day for 12 weeks
  Arms: 200mg group
Drug: Placebo matching DBPR108 tablet(100mg), Placebo matching DBPR108 tablet(50mg) — Two Placebos matching DBPR108 tablet(100mg) administered orally once a day + One Placebo matching DBPR108 tablet(50mg) administered orally once a day for 12 weeks
  Arms: placebo group

SUMMARY:
This study evaluate DRBP108 in the treatment of type 2 diabetes mellitus. The patients were randomly allocated to four groups: 50 mg, 100 mg, 200 mg and placebo group.

DETAILED DESCRIPTION:
This study was to evaluate DRBP108 in the treatment of type 2 diabetes mellitus. A total of 268 subjects were randomly allocated to four treatment arms: 50 mg, 100 mg, 200 mg or placebo group, in a 1:1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the World Health Organization(WHO) (1999) criteria for the diagnosis and classification criteria for type 2 diabetes;
* 18 ≤ age ≤ 75 years old, male or female;
* One of the following conditions:

  1. Initial diagnosis of type 2 diabetes mellitus;
  2. Patients who with type 2 diabetes diagnosed within 2 years before screening period and are treated with single-agent oral hypoglycemic agents until screening, and do not take the medicine regularly for at least 8 weeks (i.e., continuous medication for <1 week);
* 19kg/m^2 ≤ Body Mass Index（BMI ）≤ 35kg/m^2;
* 7.0% ≤ HbA1c ≤ 10.0%;
* Female subjects of childbearing age are negative in pregnancy test;
* All the subjects do not have a fertility plan during and three month after the trial;
* Subjects who fully understand the test content and possible adverse reactions and voluntarily participate in the trial and sign the informed consent form;

Exclusion Criteria:

* FPG > 15 mmol/L;
* Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg during screening period;
* Those who are known to be positive for HIV and syphilis;
* known active hepatitis B virus infection, hepatitis C virus infection;
* For patients with obvious liver diseases and chronic liver diseases, AST or ALT in screening stage was twice the normal upper limit.
* In patients with renal insufficiency, serum creatinine at screening stage was 1.5 times higher than the upper limit of normal value;
* Leukocyte and hemoglobin < lower limit of normal value, triglyceride > 5.7 mmol/L in screening stage;
* With diabetic acute complications (including diabetic ketoacidosis, hypertonic non-ketoacid diabetic coma, lactic acidosis and hypoglycemic coma), chronic complications (proliferative diabetic retinopathy, diabetic nephropathy);
* Use of insulin, pioglitazone, DPP-4 inhibitor, GLP-1 receptor agonist or any combination of two or more oral hypoglycemic drugs within 8 weeks before screening time.
* Those who need insulin therapy;
* Using and Used of glucocorticoids within 2 weeks before screening time.
* without a pacemaker, the 12-lead ECG showed II or III degree atrioventricular block, long QT syndrome or corrected QT interval （QTc）>500ms or atrial fibrillation during the screening period;
* History of epilepsy, mental illness, major depression, or previous thyroid function abnormal and still being treated, or those with organ transplants, severe chronic lung disease, and other serious heart disease, cerebrovascular disease, blood disease;
* Inflammatory bowel disease, colon ulcer, partial intestinal obstruction or chronic intestinal diseases associated with digestive and absorption diseases;
* Active pancreatitis, cholecystitis, gallstones and other digestive diseases;
* History of severe hypoglycemia;
* History of allergies with similar drugs (DPP-4 inhibitors) or those who are judged by the investigator to be allergic to the test drug;
* Pregnancy, lactating women;
* Subjects who are participating in other clinical trials or who have participated in other drug trials within 3 months prior to screening;
* Not suitable for this clinical trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
HBA1c | Baseline, week 12
  Changes in HbA1c compared to baseline at week 12

SECONDARY OUTCOMES:
HBA1c | Baseline, week 8, week4
  Changes in HbA1c compared to baseline at week 8, week 4
Fasting plasma glucose | Baseline, week 4，week 8, week 12
  Changes in Fasting plasma glucose compared to baseline at week 4,week 8, week 12
2-hour postprandial plasma glucose | Baseline, week 4，week 8, week 12
  Changes in 2-hour postprandial plasma glucose compared to baseline at week 4,week 8, week 12
fasting glucagon | Baseline, week 4，week 8, week 12
  Changes in fasting glucagon compared to baseline at week 4,week 8, week 12
fasting Insulin | Baseline, week 4，week 8, week 12
  Changes in fasting Insulin compared to baseline at week 4,week 8, week 12
active Glucagon-like peptide-1（GLP-1） | Baseline, week 4，week 8, week 12
  Changes in active（GLP-1）compared to baseline at week 4,week 8, week 12
The percentage of HbA1c≤6.5% or HbA1c≤7% | week 12
  The percentage of HbA1c≤6.5% or HbA1c≤7% at week 12
body weight | Baseline, week 4，week 8, week 12
  Changes in body weight（Kg）compared to baseline at week 4,week 8, week 12

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Peking Unversity, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang W, Yao J, Guo X, Guo Y, Yan C, Liu K, Zhang Y, Wang X, Li H, Wen Z, Wang X, Li S, Xiao X, Liu W, Li Z, Zhang L, Shao S, Ye S, Qin G, Li Y, Li F, Zhang X, Li X, Peng Y, Deng H, Xu X, Zhou L, Huang Y, Cao M, Xia X, Shi M, Dou J, Yuan J. Efficacy and safety of DBPR108 monotherapy in patients with type 2 diabetes: a 12-week, randomized, double-blind, placebo-controlled, phase II clinical trial. Curr Med Res Opin. 2020 Jul;36(7):1107-1115. doi: 10.1080/03007995.2020.1761311. Epub 2020 May 12. PMID 32338063